CLINICAL TRIAL: NCT00818701
Title: A Randomized, Double Blinded Placebo Controlled Cross-over Study of Low Dose B-type Natriuretic Peptide (Nesiritide) With or Without Concomitant Phosphodiesterase V (PDE V) Inhibition(Sildenafil) in Congestive Heart Failure Patients With Renal Dysfunction
Brief Title: Study of Low Dose Nesiritide With or Without Sildenafil in Congestive Heart Failure Patients With Renal Dysfunction
Acronym: BNP+PDEVI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: started a NIH study that is competing for same subjects
Sponsor: Mayo Clinic (Other)
Responsible Party: Dr Horng H. Chen, Mayo Clinc
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 08-004797; BNP + PDEVI
Record Dates: First submitted 2009-01-06; First posted 2009-01-08 (Estimated); Last update posted 2010-09-24 (Estimated); Status verified 2010-09

CONDITIONS: Congestive Heart Failure; Renal Dysfunction
Keywords: Congestive Heart Failure; Congestive Heart Failure with a NYHF Class 2-3; Ejection Fraction of 35 or less
MeSH Terms: conditions — Heart Failure; Renal Insufficiency | interventions — Natriuretic Peptide, Brain; Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: low dose BNP alone (Placebo Comparator): low dose BNP with placebo
  Interventions: Drug: low dose Nesiritide
- 2: low dose BNP + PDEVI (Active Comparator): low dose BNpo + PDEVI
  Interventions: Drug: nesiritide, Sildenafil

INTERVENTIONS:
Drug: low dose Nesiritide — Nesiritide infusion 0.005ug/kg/min
  Other Names: Natracor
  Arms: 1: low dose BNP alone
Drug: nesiritide, Sildenafil — Nesiritide 0.005ug/kg/min Sildenafil 50 mg
  Other Names: Natrecor; Viagra
  Arms: 2: low dose BNP + PDEVI

SUMMARY:
The purpose of the study is to show that low dose recombinant BNP coupled with phosphodiesterase V inhibition will improve renal dysfunction and promote relief of volume overload in patinets with acute decompensated heart failure complicated by the cardiorenal syndrome.

DETAILED DESCRIPTION:
Renal dysfunction is a common comorbidity, as well as a common and progressive complication, of heart failure (HF). Increasingly, the clinical syndrome of HF is one of "cardiorenal" failure owing to the frequent presentation of combined cardiac and renal dysfunction. Recent studies have established the prognostic importance of renal dysfunction in patients with chronic HF. An analysis of the patients in the second prospective randomized study of Ibopamine on mortality and efficacy (PRIME) by Hillege et al1 demonstrated that estimated glomerular filtration rate (GFR) is the most powerful predictor of mortality, exceeding functional status and ejection fraction (EF).

In an ongoing prospective study, we are assessing the neurohumoral and renal hemodynamic profile of hospitalized patients with ADHF who do or do not develop the CRS. Our preliminary findings suggest that indeed the combination of pronounced activation of renin-angiotensin-aldosterone system (RAAS), decreased renal perfusion pressure and importantly, a relative deficiency of the natriuretic peptides (despite marked volume overload) predisposes to the development of CRS.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction 35% assessed by echocardiography, nuclear scan or left ventriculogram within the past 2 years
* Stable (NYHA) class II and III symptoms as defined by:

  1. no change in NYHA symptoms over the past 3 months;
  2. on stable doses of ACE inhibitor and beta blocker for one month;
  3. no episode of decompensated CHF over the past 3 months.
* Calculated creatinine clearance of equal or less than 60 ml/min and greater than 30 ml/min, using the Cockcroft-Gault formula assessed within the past 12 months

Exclusion Criteria:

* Nitrates or alpha blockers
* Prior diagnosis of intrinsic renal diseases including renal artery stenosis of > 50%
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Hospitalization for decompensated CHF during the past 3 months
* Myocardial infarction within 3 months of screening
* Unstable angina within 3 months of screening or any evidence of myocardial ischemia
* Significant valvular stenosis, hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening or other evidence of significantly compromised CNS perfusion
* Serum sodium of < 125 mEq/dL or > 150 mEq/dL
* Serum potassium of < 3.5 mEq/dL or > 5.7 mEq/dL
* Hemoglobin < 10 gm/dl
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* Received an investigational drug within 1 month prior to dosing
* Patients with an allergy to iodine.
* Female subject who is pregnant or breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To determine the efficacy of low dose BNP alone vs low dose BNP + PDE V inhibition in improving renal function in patients with CHF and renal dysfunction. (Calculated creatinine clearance = or < than 60 ml/min and > 30 ml/min, within 12 months.) | prospective

SECONDARY OUTCOMES:
We also want to characterize both plasma and urinary humoral profile in these patients. | prospective

CONTACTS AND LOCATIONS:
Overall Officials: Horng H Chen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States